CLINICAL TRIAL: NCT04429594
Title: Study of the Incidence of SARS-CoV-2 Infection in the Alpes-Maritimes Department by Analysis of the Specific Humoral and Cellular Response During Deconfinement
Brief Title: Study of the Incidence of SARS-CoV-2 Infection (COVID-19)
Acronym: CovImmune 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-PP-14
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Coronavirus Infections
MeSH Terms: conditions — Coronavirus Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- volonteers (Other)
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — blood sampling at J0, M6, M12, M24, M36, M48, M60

SUMMARY:
This is a prospective observational cohort study that will define the prevalence and incidence of CA-SARS-Cov2 infection using serological and PCR tests in a group of subjects during deconfinement. The team wishes to include approximately 1000 subjects in this study.

The health crisis through containment has also created unprecedented environmental conditions with the very clear decrease in economic activities and a consequent decrease in exposure to the main air pollutants. The aim is therefore to carry out a case-control study in which each subject will be his or her own control in unexposed condition (to PM2.5, PM10, NO...) then exposed (after the recovery of economic activity and the usual levels of air pollutants) and to measure the impact of these pollutants on the immune system and epigenetic markers taking into account seasonality.

The occurrence of infectious, cardiovascular, allergic and autoimmune events will then be measured according to the immunological profiles measured at inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Any major subject, voluntary, exposed to the public from 11 May 2020 informed of the study by partner institutions (Departmental Council 06), affiliated to a social security scheme,

Exclusion Criteria:

* Subject protected by law under tutorship or guardianship, or who cannot participate in a clinical study under the terms of Article L. 1121-16 of the French Public Health Code

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-07-28 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
positive serologies | 12 months
  number of positive serologies

CONTACTS AND LOCATIONS:
Locations (1):
- University Nice Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Graca D, Brglez V, Allouche J, Zorzi K, Fernandez C, Teisseyre M, Cremoni M, Benzaken S, Pradier C, Seitz-Polski B. Both Humoral and Cellular Immune Responses to SARS-CoV-2 Are Essential to Prevent Infection: a Prospective Study in a Working Vaccinated Population from Southern France. J Clin Immunol. 2023 Nov;43(8):1724-1739. doi: 10.1007/s10875-023-01558-9. Epub 2023 Aug 22. PMID 37606852
- [Derived] Buscot M, Cremoni M, Graca D, Brglez V, Courjon J, Allouche J, Teisseyre M, Boyer L, Barriere J, Chamorey E, Carles M, Seitz-Polski B. Breakthrough infections due to SARS-CoV-2 Delta variant: relation to humoral and cellular vaccine responses. Front Immunol. 2023 Mar 30;14:1145652. doi: 10.3389/fimmu.2023.1145652. eCollection 2023. PMID 37063916